CLINICAL TRIAL: NCT03219879
Title: Telephone-administered Cognitive-behavioral Relapse Prevention for Patients with Chronic and Recurrent Depression: a Multi-center Randomized Clinical Trial
Brief Title: Telephone-administered Relapse Prevention for Depression
Acronym: NaTel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100019_166009 / 1
Record Dates: First submitted 2017-06-20; First posted 2017-07-18 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Depressive Disorder
Keywords: Relapse prevention; Persistent depressive disorder; Recurrent depressive disorder; Telephone-based intervention; Cognitive behavioral therapy
MeSH Terms: conditions — Depressive Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telephone-administered continuation therapy (Experimental): Cognitive-behavioral continuation therapy (T-CT) delivered over the telephone by trained psychotherapist
  Interventions: Behavioral: Telephone-administered continuation therapy
- Usual care (Active Comparator): Treatment as usual
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Telephone-administered continuation therapy — The intervention includes eight therapy sessions of approx. 50 minutes duration delivered over the telephone by trained psychotherapists over a time period of six months. The intervention is grounded in the principles of psychological continuation therapy and relapse prevention, and includes strategies such as transferring helpful elements of acute-phase cognitive-behavioral therapy (CBT) for depression to daily life. T-CT is offered in addition to usual care.
  Arms: Telephone-administered continuation therapy
Other: Usual care — Usual care without any study-related intervention
  Other Names: Treatment as usual (TAU)
  Arms: Usual care

SUMMARY:
This study determines the effectiveness of telephone-delivered cognitive-behavioral continuation therapy (T-CT) in comparison to usual care in people with recurrent or chronic depression. The primary research question is whether participating in T-CT reduces depressive relapses. The continuation therapy comprises eight therapy sessions delivered over the telephone by a trained therapist over a period of approximately six months following acute-phase psychotherapy.

DETAILED DESCRIPTION:
Major depression is a serious mental disorder that often takes a recurrent or chronic course causing enduring individual suffering as well as immense direct and indirect health costs. Research indicates that psychological continuation interventions following successful acute-phase therapy are effective in preventing depressive relapse and recurrence but access to these interventions is limited. Systematic psychological continuation interventions are hardly implemented in health care yet, and research shows that there are obstacles concerning access to and compliance for these interventions in a face-to-face setting underlining the need for alternative ways of delivery. The present study ("NaTel study") aims to investigate the effectiveness of telephone-administered cognitive-behavioral continuation therapy (T-CT) following acute-phase psychotherapy. The primary research question is whether participating in T-CT reduces depressive relapses within an observation period of 18 months compared with usual care alone. T-CT comprises eight therapy sessions delivered over the telephone by a trained therapist over a period of approximately six months after acute-phase therapy. Focus of the structured intervention is to train and foster relapse prevention strategies and to facilitate the transfer of skills acquired during acute-phase therapy to daily life. The effectiveness of T-CT as add-on to usual care is tested in a two-parallel group, multicenter, evaluator-blind clinical trial in patients with chronic/persistent or recurrent depressive disorder. Upon acute-phase therapy termination patients who have responded to cognitive behavioral therapy are randomized either to T-CT or usual care alone. Primary outcome of this study is relapse of a depressive episode. Relapse is determined by investigators blind to the study conditions based on clinical interviews conducted at months 6, 12, and 18 of follow-up. Further secondary outcome criteria are assessed with interviews and self-report questionnaires at various time points during follow-up. Overall, the study lasts approximately 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent major depressive disorder or chronic/persistent depressive disorder based on the criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), or first major depressive episode with an elevated risk for relapse (defined as the presence of at least of the following clinical characteristics: index episode duration ≥ six months; severity of the index episode at least moderate; DSM-5 comorbidity; residual symptoms at the end of index treatment)
* Having regularly terminated acute-phase CBT for depression (index treatment)
* Having achieved therapeutic response during index therapy defined as at least 25%-improvement in depressive symptoms between start and end of acute-phase therapy based on a standardized symptom measure (e.g. PHQ-9, or Beck Depression Inventory; BDI)
* Having experienced partial or full remission at the end of the index treatment based on DSM-5 criteria for major depressive disorder
* Sufficient command of German language
* Having given written informed consent

Exclusion Criteria:

* Unstable psychopharmacological medication regimen (either with or without antidepressant (AD) medication) at the end of the index treatment, i.e. change in type or dosage of medication envisaged at the end of index treatment
* Acute risk for suicide based on clinical practice guidelines; patients with self-reported suicidal ideation are eligible as long as the treatment is deemed safe by the clinician's judgment
* A history of or acute psychotic symptoms, bipolar disorder, or organic brain disorder
* Severe cognitive impairment based on clinical evaluation during index treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2023-04-08 (Actual); Study Completion 2023-04-08 (Actual)

PRIMARY OUTCOMES:
Relapse of a major depressive episode | 6 months, 12 months, and 18 months after baseline
  Relapse is assessed with the Longitudinal Interval Follow-up Evaluation (LIFE) and defined as a Psychiatric Status Rating (PSR) of PSR=5 or PSR=6 on the 6-point PSR scale for affective disorders for at least two consecutive weeks during a total of 18 months follow-up according to evaluators who are blinded to group allocation

SECONDARY OUTCOMES:
Well-weeks | 6 months, 12 months, and 18 months after baseline
  Number of weeks without depressive symptoms defined as weeks with a PSR=1 or PSR=2 on the PSR 6-point scale for affective disorders assessed with the LIFE at month 6, 12 and 18 of follow-up according to blind evaluators
Depressive symptoms | Baseline, 3 months, 6 months, and 12 months after baseline
  Self-reported depressive symptoms assessed with the Patient Health Questionnaire-9 (PHQ-9) at baseline, 3-, 6-, and 12-month follow-up
Health-related quality of life | Baseline, 3 months, 6 months, and 12 months after baseline
  Health-related quality of life (HrQoL) based on patient self-report assessed with the 12-Item Short Form Health Survey (SF-12) at baseline, 3-, 6- and12-month follow-up
Anxiety symptoms | Baseline, 3 months, 6 months, and 12 months after baseline
  Self-reported anxiety symptoms assessed with the General Anxiety Disorder 7 (GAD-7) screener at baseline, 3-, 6-, and 12-month follow-up
Psychosocial functioning | 6 months and 12 months after baseline
  Psychosocial functioning assessed with the LIFE-Range of Impaired Functioning Tool (LIFE-RIFT) and Global Assessment of Functioning (GAF) based on monthly ratings by blind evaluators
Cost of health care utilization | Baseline, 6 months, and 12 months after baseline
  Direct and indirect cost derived from health care utilization and productivity loss are assessed with the Client Sociodemographic and Service Receipt Inventory (CSSRI-D) at baseline, 6- and 12-month follow-up
Cost-effectiveness | Baseline, 6 months, and 12 months after baseline
  Health-related quality of life assessments for health economic analyses by the determination of Quality-Adjusted Life Years (QALYs) are based on the EuroQol-five dimension questionnaire five-level version (EQ-5D-5L) administered at baseline, 6- and 12-month follow-up

OTHER OUTCOMES:
T-CT acceptability | 6 months after baseline
  Satisfaction with and acceptability of the telephone-intervention from therapist and participant perspective at 6-month follow-up (T-CT group only) assessed with a customized self-report evaluation questionnaire
Treatment satisfaction | Baseline, and 6 months after baseline
  General treatment satisfaction from participant perspective assessed with Client Satisfaction Questionnaire (ZUF-8) at baseline (both groups) and 6-month follow-up (T-CT group only)
Self-confidence | Baseline, 6 months, and 12 months after baseline
  Participants' self-reported general levels of confidence assessed at baseline, 6- and 12-month follow-up
Physical activity | Baseline, 6 months, and 12 months after baseline
  Participants' levels of physical activity assessed with the International Physical Activity Questionnaire Short Form (IPAC-SF) at baseline, 6- and 12-month follow-up
Self-efficacy for depression self-management | Baseline, 3 months, 6 months, and 12 months after baseline
  Self-efficacy for depression self-management assessed via self-report questionnaire at baseline, 3-, 6- and 12-month follow-up
Self-management behaviors | Baseline, 3 months, 6 months, and 12 months after baseline
  Depression-related self-management behaviors assessed via self-report questionnaire at baseline, 3-, 6-, and 12-month follow-up
Interpersonal emotion regulation skills | Baseline, 6 months, and 12 months after baseline
  Participants' interpersonal emotion regulation skills assessed with the Interpersonal Emotion Regulation Questionnaire (IERQ) at baseline, 6- and 12-month follow-up
Therapeutic alliance | Baseline, 3 months, and 6 months after baseline
  Therapeutic alliance assessed with the Working Alliance Questionnaire-short revised (WAI-SR) from therapist and participant perspective assessed at baseline (both groups), as well as 3- and 6-month follow-up (T-CT group only)

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Watzke, Prof, Principal Investigator — University of Zurich; Markus Wolf, PhD, Principal Investigator — University of Zurich
Locations (11):
- Institut für Klinische Psychologie, Krankenhaus Bad Cannstatt, Klinikum Stuttgart, Stuttgart, Germany
- Switzerland (10):
  - Universitätsklinik für Psychiatrie und Psychotherapie, Universität Bern, Bern
  - Zentrum Psychiatrie und Psychotherapie stationär, Psychiatrische Dienste Aargau AG, Brugg
  - Zentrum für Psychiatrie und Psychotherapie, Klinik Gais AG, Gais
  - Klinik für Psychiatrie und Psychotherapie, Psychiatrisches Zentrum AR, Herisau
  - Klinik SGM Langenthal, Langenthal
  - Zentrum für seelische Gesundheit, Privatklinik Meiringen, Meiringen
  - Zentrum für Psychiatrie und Psychotherapie Klinik Zugersee, Triaplus AG, Oberwil
  - Psychiatrische und Psychotherapeutische Spezialklinik für Frauen, Klinik Meissenberg AG, Zug
  - Klinik für Psychiatrie und Psychotherapie, UniversitätsSpital Zürich, Zurich
  - Praxisstelle Psychotherapie, Universität Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Brief abstract of the trial — http://www.psychologie.uzh.ch/de/fachrichtungen/klipfor/forschung/forschungsprojekte.html